CLINICAL TRIAL: NCT02813135
Title: European Proof-of-Concept Therapeutic Stratification Trial of Molecular Anomalies in Relapsed or Refractory Tumors
Acronym: ESMART
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government); Fight Kids Cancer (Other); Fondation ARC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-000133-40; 2016/2396 (Other: CSET Number); 2024-514791-40-00 (EU CTIS Number)
Record Dates: First submitted 2016-06-16; First posted 2016-06-24 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cancer
Keywords: Children; Adolescents; Young adults; Recurrent malignancies; Refractory malignancies
MeSH Terms: conditions — Neoplasms | interventions — ribociclib; Topotecan; Temozolomide; Everolimus; adavosertib; Carboplatin; olaparib; Irinotecan; vistusertib; Nivolumab; Cyclophosphamide; AZD 6244; enasidenib; lirilumab; CYC065; Cytarabine; Dexamethasone; Calcium Dobesilate; ceralasertib; futibatinib; capmatinib; avelumab; peposertib; capivasertib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- Arm A. Ribociclib + Topotecan and Temozolomide (Experimental): Topotecan iv QD and temozolomide capsules orally QD Days 1 to 5; Ribociclib capsules or oral solution orally QD from Day 6 to 20 of a 28 day cycle.
  Interventions: Drug: Ribociclib; Drug: Topotecan; Drug: Temozolomide
- Arm B. Ribociclib + Everolimus (Experimental): Ribociclib capsules or oral solution orally QD for 21 days of each 28 day cycle; Everolimus orodispersible tablets orally QD for 28 days.
  Interventions: Drug: Ribociclib; Drug: Everolimus
- ARM C. Adavosertib + Carboplatin (Experimental): Adavosertib capsules orally BID 3 days on / 4 days off in week 1; Carboplatin iv QD AUC 5 on Day 1 of a 21 day cycle.
  Interventions: Drug: Adavosertib; Drug: Carboplatin
- Arm D. Olaparib + Irinotecan (Experimental): Olaparib tablets orally BID on Day 1-10 of a 21 day cycle Irinotecan iv QD on Day 4-8 of a 21 day cycle.
  Interventions: Drug: Olaparib; Drug: Irinotecan
- Arm E. Vistusertib single agent (Experimental): Vistusertib tablets orally BID 2 days on/5 days off per week of a 28 day cycle.
  Interventions: Drug: Vistusertib
- Arm F. Vistusertib + Topotecan and Temozolomide (Experimental): Topotecan iv QD and temozolomide capsules orally QD Days 1 to 5; Vistusertib tablets orally BID 3 days on/4 days off per week of a 28 day cycle.
  Interventions: Drug: Topotecan; Drug: Temozolomide; Drug: Vistusertib
- Arm G. Nivolumab + Cyclophosphamide +/- Radiotherapy (Experimental): Nivolumab iv QD every 2 weeks of a 28 day cycle (Days 1 and 15); Cyclophosphamide tablets or oral solution orally BID, 1 week on/1 week off; Palliative irradiation/radiofrequency/cryotherapy starting 2 weeks after the first nivolumab injection.
  Interventions: Drug: Nivolumab; Drug: Cyclophosphamide
- Arm H. Selumetinib + Vistusertib (Experimental): Selumetinib capsules twice daily on a continous administration. Vistusertib orally twice daily on an intermittent schedule : 2 days on / 5 days off per week of a 28 day cycle.
  Interventions: Drug: Vistusertib; Drug: Selumetinib
- Arm I. Enasidenib (Experimental): Enasidenib tablets or sprinkle solution orally on a continuous dosing once daily (QD) per 28 day cycle.
  Interventions: Drug: Enasidenib
- Arm J. Lirilumab + Nivolumab (Experimental): Nivolumab iv QD on Day 1 and 15 of a 28 day cycle; Lirilumab iv QD on Day 1 of a 28 day cycle
  Interventions: Drug: Nivolumab; Drug: Lirilumab
- Arm K. Fadraciclib (CYC065) + Temozolomide (Experimental): Fadraciclib iv QD on Day 1 (+/- 15) of a 28 day cycle Temozolomide capsules orally QD on Day 1-5 of a 28 day cycle
  Interventions: Drug: Temozolomide; Drug: Fadraciclib
- Arm L. Fadraciclib (CYC065) + Cytarabine (Experimental): Fadraciclib iv QD on Day 1 (+/- 15) of a 28 day cycle Cytarabine iv or sc on Day 2-5 and Day 8-11 of a 28 day cycle
  Interventions: Drug: Fadraciclib; Drug: Cytarabine
- Arm M. Ribociclib + Everolimus +/- Dexamethasone (Experimental): Ribociclib capsules or tablets orally QD on Day 1-21 of a 28 day cycle. Everolimus dispersible tablets orally QD on a continuous dosing per 28 day cycle.
  For patients with leukemia and lymphoma:
  Dexamethasone orally or iv on Day 1-7 of each 28 day cycle. For patients with ALL, AML and Non-Hodgkin Lymphoma (NHL), Intrathecal chemotherapy will be administered additionally as per standard practice depending on CNS status.
  Interventions: Drug: Ribociclib; Drug: Everolimus; Drug: Dexamethasone
- Arm N. Ceralasertib (AZD6738) + Olaparib (Experimental): Olaparib tablets orally BID per 28 days Ceralasertib tablets QD or BID per 28 day cycle
  Interventions: Drug: Olaparib; Drug: Ceralasertib
- Arm O. Futibatinib (TAS-120) (Experimental): Futibatinib tablets orally on a continuous dosing QD per 28 day cycle
  Interventions: Drug: Futibatinib
- Arm P. Capmatinib (INC280) + Everolimus (Experimental): Capmatinib tablets orally on a continuous dosing BID per 28 day cycle. Everolimus dispersible tablets orally QD on a continuous dosing per 28 day cycle.
  Interventions: Drug: Everolimus; Drug: Capmatinib
- Arm Q. Peposertib + Avelumab and Metronomic Temozolomide (Experimental): Peposertib tablets orally on a continuous dosing BID per 28 day cycle Avelumab IV QD on Day 1 and Day 15 of a 28 day cycle Temozolomide capsules orally QD 5 days/week of a 28 day cycle
  Interventions: Drug: Temozolomide; Drug: Avelumab; Drug: Peposertib
- Arm R. Capivasertib + metronomic Vinorelbine (Experimental): Capivasertib tablets orally BID on Day 1-4/week (4 days on/3 days off, every week) of a 28 day cycle.
  Vinorelbine soft capsules orally once daily on Day 1, 3 and 5/week of a 28 day cycle.
  Interventions: Drug: Capivasertib; Drug: Vinorelbine

INTERVENTIONS:
Drug: Ribociclib
  Other Names: Kisqali; LEE011
  Arms: Arm A. Ribociclib + Topotecan and Temozolomide; Arm B. Ribociclib + Everolimus; Arm M. Ribociclib + Everolimus +/- Dexamethasone
Drug: Topotecan
  Other Names: Hycamtin
  Arms: Arm A. Ribociclib + Topotecan and Temozolomide; Arm F. Vistusertib + Topotecan and Temozolomide
Drug: Temozolomide
  Other Names: Temodar
  Arms: Arm A. Ribociclib + Topotecan and Temozolomide; Arm F. Vistusertib + Topotecan and Temozolomide; Arm K. Fadraciclib (CYC065) + Temozolomide; Arm Q. Peposertib + Avelumab and Metronomic Temozolomide
Drug: Everolimus
  Other Names: Afinitor; votubia
  Arms: Arm B. Ribociclib + Everolimus; Arm M. Ribociclib + Everolimus +/- Dexamethasone; Arm P. Capmatinib (INC280) + Everolimus
Drug: Adavosertib
  Other Names: AZD1775
  Arms: ARM C. Adavosertib + Carboplatin
Drug: Carboplatin
  Other Names: Paraplatin
  Arms: ARM C. Adavosertib + Carboplatin
Drug: Olaparib
  Other Names: Lynparza
  Arms: Arm D. Olaparib + Irinotecan; Arm N. Ceralasertib (AZD6738) + Olaparib
Drug: Irinotecan
  Other Names: Camptosar; CPT-11
  Arms: Arm D. Olaparib + Irinotecan
Drug: Vistusertib
  Other Names: AZD2014
  Arms: Arm E. Vistusertib single agent; Arm F. Vistusertib + Topotecan and Temozolomide; Arm H. Selumetinib + Vistusertib
Drug: Nivolumab
  Other Names: Opdivo
  Arms: Arm G. Nivolumab + Cyclophosphamide +/- Radiotherapy; Arm J. Lirilumab + Nivolumab
Drug: Cyclophosphamide
  Other Names: Cytoxan
  Arms: Arm G. Nivolumab + Cyclophosphamide +/- Radiotherapy
Drug: Selumetinib
  Other Names: Koselugo
  Arms: Arm H. Selumetinib + Vistusertib
Drug: Enasidenib
  Other Names: Idhifa
  Arms: Arm I. Enasidenib
Drug: Lirilumab
  Other Names: BMS-986015
  Arms: Arm J. Lirilumab + Nivolumab
Drug: Fadraciclib
  Other Names: CYC065
  Arms: Arm K. Fadraciclib (CYC065) + Temozolomide; Arm L. Fadraciclib (CYC065) + Cytarabine
Drug: Cytarabine
  Other Names: Arabinosylcytosine; Cytosar-U
  Arms: Arm L. Fadraciclib (CYC065) + Cytarabine
Drug: Dexamethasone
  Other Names: Decadron; Dexasone; Diodex; Hexadrol; Maxidex
  Arms: Arm M. Ribociclib + Everolimus +/- Dexamethasone
Drug: Ceralasertib
  Other Names: AZD6738
  Arms: Arm N. Ceralasertib (AZD6738) + Olaparib
Drug: Futibatinib
  Other Names: Tas-120
  Arms: Arm O. Futibatinib (TAS-120)
Drug: Capmatinib
  Other Names: Tabrecta; INC280
  Arms: Arm P. Capmatinib (INC280) + Everolimus
Drug: Avelumab
  Other Names: BAVENCIO
  Arms: Arm Q. Peposertib + Avelumab and Metronomic Temozolomide
Drug: Peposertib
  Arms: Arm Q. Peposertib + Avelumab and Metronomic Temozolomide
Drug: Capivasertib
  Other Names: TRUQAP; AZD5363
  Arms: Arm R. Capivasertib + metronomic Vinorelbine
Drug: Vinorelbine
  Other Names: Navelbine
  Arms: Arm R. Capivasertib + metronomic Vinorelbine

SUMMARY:
This proof-of-concept platform trial is designed to cover the targeting of several survival pathways in oncogenesis that are currently not adequately employed for pediatric patients in Europe (Geoerger 2017; Geoerger 2019).

The aims of the trial are:

1. To determine the recommended phase II dose (RP2D) of a specific anticancer agent and/or a relevant combination in a pediatric population, to document its tolerability and
2. To explore first signals of activity in a molecularly enriched study population.

DETAILED DESCRIPTION:
The first molecular profiling protocols have been launched in Europe (MOSCATO-01 (Geoerger 2014), MAPPYACTS, INFORM, iTHER, SM-PAEDS, etc.) determining multiple actionable alterations in pediatric recurrent cancers. Increasingly, stratified approaches are being implemented to enrich clinical trials of molecularly targeted agents and possibly improve outcomes in specific populations i.e. a molecularly enriched/predictive biomarker-driven approach. The diversity and heterogeneity of the detected molecular alterations and the low number of pediatric patients mandate an adapted, innovative trial design for the attributed treatment options in order to satisfy the current unmet medical need.

This basket trial is designed to cover the targeting of several survival pathways in oncogenesis that are currently not adequately employed for pediatric patients in Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be diagnosed with a haematologic or solid tumor malignancy that has progressed despite standard therapy, or for which no effective standard therapy exists.
2. Age < 18 years at inclusion; patients 18 years and older may be included after discussion with the sponsor if they have a pediatric recurrent/refractory malignancy.
3. Patient must have had advanced molecular profiling (i.e. WES/WGS +/- RNAseq) of their recurrent or refractory tumor i.e. at the time of disease progression/relapse; exceptionally patients with advanced molecular profiling at diagnosis may be allowed.
4. Evaluable or measurable disease as defined by standard imaging criteria for the patient's tumor type (RECIST v1.1, RANO criteria for patients with HGG, INRC criteria for patients with NB, Leukemia criteria, etc.).
5. Patients with relapsed or refractory leukemia are eligible for this study.
6. Performance status: Karnofsky performance status (for patients >12 years of age) or Lansky Play score (for patients ≤12 years of age) ≥ 70%. Patients who are unable to walk because of paralysis or stable neurological disability, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
7. Life expectancy ≥ 3 months
8. Adequate organ function:

   Hematologic criteria (Leukemia patients are excluded from hematological criteria):
   * Peripheral absolute neutrophil count (ANC) ≥ 1000/μL(unsupported)
   * Platelet count ≥ 100,000/μL (unsupported)
   * Hemoglobin ≥ 8.0 g/dL (transfusion is allowed)

   Cardiac function:
   * Shortening fraction (SF) >29% (>35% for children < 3 years) and left ventricular ejection fraction (LVEF) ≥50% at baseline, as determined by echocardiography (mandatory only for patients who have received cardiotoxic therapy).
   * Absence of QTc prolongation (QTc > 450 msec on baseline ECG, using the Fridericia correction [QTcF formula]) or other clinically significant ventricular or atrial arrhythmia.

   Renal and hepatic function:
   * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) for age
   * Total bilirubin ≤ 1.5 x ULN
   * Alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≤ 2,5 x ULN; aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase/SGOT ≤ 2,5 x ULN except in patients with documented tumor involvement of the liver who must have AST/SGOT and ALT/SGPT ≤ 5 x ULN.
9. Able to comply with scheduled follow-up and with management of toxicity.
10. Females of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to initiation of treatment. Sexually active women of childbearing potential must agree to use acceptable and appropriate contraception during the study and for at least 6 months after the last study treatment administration. Sexually active males patients must agree to use condom during the study and for at least 6 months (7 months for arm J) after the last study treatment administration. Acceptable contraception are defined in CTFG Guidelines "Recommendations related to contraception and pregnancy testing in clinical trials"
11. For all oral medications patients must be able to comfortably swallow capsules (except for those for which an oral solution is available); nasogastric or gastrostomy feeding tube administration is allowed only if indicated.
12. Written informed consent from parents/legal representative, patient, and age-appropriate assent before any study-specific screening procedures are conducted according to local, regional or national guidelines.
13. Patient affiliated to a social security regimen or beneficiary of the same according to local requirements.

Exclusion Criteria:

1. Patients with symptomatic central nervous system (CNS) metastases who are neurologically unstable or require increasing doses of corticosteroids or local CNS-directed therapy to control their CNS disease. Patients on stable doses of corticosteroids for at least 7 days prior to receiving study drug may be included.
2. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter drug absorption of oral drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome).
3. Clinically significant, uncontrolled heart disease (including history of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality, unstable ischemia,congestive heart failure within 12 months of screening)
4. Active viral hepatitis or known human immunodeficiency virus (HIV) infection or any other uncontrolled infection.
5. Presence of any ≥ CTCAE grade 2 treatment-related toxicity with the exception of alopecia, ototoxicity or peripheral neuropathy.
6. Systemic anticancer therapy within 21 days of the first study dose or 5 times its half-life, whichever is less.
7. Previous myeloablative therapy with autologous hematopoietic stem cell rescue within 8 weeks of the first study drug dose
8. Allogeneic stem cell transplant within 3 months prior to the first study drug dose. Patients receiving any agent to treat or prevent graft-versus host disease (GVHD) post bone marrow transplant are not eligible for this trial.
9. Radiotherapy (non-palliative) within 21 days prior to the first dose of drug (or within 6 weeks for therapeutic doses of MIBG or craniospinal irradiation).
10. Major surgery within 21 days of the first dose. Gastrostomy, ventriculo-peritoneal shunt, endoscopic ventriculostomy, tumor biopsy and insertion of central venous access devices are not considered major surgery, but for these procedures, a 48 hour interval must be maintained before the first dose of the investigational drug is administered.
11. Currently taking medications with a known risk of prolonging the QT interval or inducing Torsades de Pointes (Refer to Appendix 8).
12. Currently taking medications that are mainly metabolized by CYP3A4/5, CYP2C8, CYP2C9, CYP2C19, CYP2D6 or the drug transporters Pgp (MDR1), BCRP, OATP1B1, OATP1B3, OCT1 and OCT2 and have a low therapeutic index that cannot be discontinued at least 7 days or 5 x reported elimination half-life prior to start of treatment with any of the investigational drugs and for the duration of the study (Refer to Appendix 9).
13. Known hypersensitivity to any study drug or component of the formulation.
14. Pregnant or nursing (lactating) females.
15. Vaccinated with live, attenuated vaccines within 4 weeks of the first dose of study drug.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 472 (Estimated)
Dates: Start 2016-08-03 (Actual); Primary Completion 2031-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) | During the first cycle
  Defined as the adult recommended dose (adjusted for weight or BSA) if toxicity and/or PK profiling are similar in children and in adults, or a higher dose, providing it is below or equal to the maximum tolerated dose (MTD)
Maximum Tolerated Dose (MTD) | During the first cycle
  The MTD will be defined as the dose associated with or closest to 25% of Dose Limiting Toxicities (DLTs)
Objective Response Rate (ORR) | During treatment period
  Defined as the proportion of participants who achieved a confirmed complete response (CR) or partial response (PR) assessed by investigators.
  In patients with leukemia, ORR is defined as the percentage of patients attaining CR, CRi or CRp.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | Depending on the treatment arm
  To characterize single or multiple-dose PK of the agent(s)
Progression Free Survival (PFS) | From treatment initiation until the date of first documented progression or death
  Defined as the time from treatment initiation until the date of first documented progression (clinically or radiologically) or death from any cause. Patients alive and free of progression at the cut-off date will be censored at the last assessment date.
Evaluation of duration of response (DoR) | Between the first document response and the time of first documented progression
  Defined as the time period between the first documented response (complete response (CR) or partial response (PR)) and the time of progression, according to RECIST v1.1, RANO criteria for patients with HGG, INRC criteria for patients with NB, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Geoerger, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (21):
- Rigshospitalet, Copenhagen, Denmark
- France (9):
  - Gustave Roussy, Villejuif, Val De Marne
  - CHU Angers, Angers
  - CHU Pellegrin, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital de La Timone, Marseille
  - CHU Nantes, Nantes
  - Institut Curie, Paris
  - Hôpital Armand Trousseau, Paris
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Ospedale Infantile Regina Margherita, Torino
- Prinses Maxima Centrum, Utrecht, Netherlands
- Spain (3):
  - Vall d'Hebron, Barcelona
  - Hospital del Nino Jesus, Madrid
  - Hospital Universitario La Fe, Valencia
- United Kingdom (5):
  - Birmingham Children's Hospital, Birmingham
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle
  - Pediatric and Adolescent Oncology The Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berlanga P, Pierron G, Lacroix L, Chicard M, Adam de Beaumais T, Marchais A, Harttrampf AC, Iddir Y, Larive A, Soriano Fernandez A, Hezam I, Chevassus C, Bernard V, Cotteret S, Scoazec JY, Gauthier A, Abbou S, Corradini N, Andre N, Aerts I, Thebaud E, Casanova M, Owens C, Hladun-Alvaro R, Michiels S, Delattre O, Vassal G, Schleiermacher G, Geoerger B. The European MAPPYACTS Trial: Precision Medicine Program in Pediatric and Adolescent Patients with Recurrent Malignancies. Cancer Discov. 2022 May 2;12(5):1266-1281. doi: 10.1158/2159-8290.CD-21-1136. PMID 35292802
- [Derived] Morscher RJ, Brard C, Berlanga P, Marshall LV, Andre N, Rubino J, Aerts I, De Carli E, Corradini N, Nebchi S, Paoletti X, Mortimer P, Lacroix L, Pierron G, Schleiermacher G, Vassal G, Geoerger B. First-in-child phase I/II study of the dual mTORC1/2 inhibitor vistusertib (AZD2014) as monotherapy and in combination with topotecan-temozolomide in children with advanced malignancies: arms E and F of the AcSe-ESMART trial. Eur J Cancer. 2021 Nov;157:268-277. doi: 10.1016/j.ejca.2021.08.010. Epub 2021 Sep 17. PMID 34543871
- [Derived] Bautista F, Paoletti X, Rubino J, Brard C, Rezai K, Nebchi S, Andre N, Aerts I, De Carli E, van Eijkelenburg N, Thebaud E, Corradini N, Defachelles AS, Ducassou S, Morscher RJ, Vassal G, Geoerger B. Phase I or II Study of Ribociclib in Combination With Topotecan-Temozolomide or Everolimus in Children With Advanced Malignancies: Arms A and B of the AcSe-ESMART Trial. J Clin Oncol. 2021 Nov 10;39(32):3546-3560. doi: 10.1200/JCO.21.01152. Epub 2021 Aug 4. PMID 34347542
- [Derived] Pasqualini C, Rubino J, Brard C, Cassard L, Andre N, Rondof W, Scoazec JY, Marchais A, Nebchi S, Boselli L, Grivel J, Aerts I, Thebaud E, Paoletti X, Minard-Colin V, Vassal G, Geoerger B. Phase II and biomarker study of programmed cell death protein 1 inhibitor nivolumab and metronomic cyclophosphamide in paediatric relapsed/refractory solid tumours: Arm G of AcSe-ESMART, a trial of the European Innovative Therapies for Children With Cancer Consortium. Eur J Cancer. 2021 Jun;150:53-62. doi: 10.1016/j.ejca.2021.03.032. Epub 2021 Apr 20. PMID 33892407
- [Derived] Rossoni C, Bardet A, Geoerger B, Paoletti X. Sequential or combined designs for Phase I/II clinical trials? A simulation study. Clin Trials. 2019 Dec;16(6):635-644. doi: 10.1177/1740774519872702. Epub 2019 Sep 20. PMID 31538815